CLINICAL TRIAL: NCT02490280
Title: Examining Biomarkers of Anxiety in a Healthy Sample of Youth and Adults
Brief Title: Examining Cortisol and Alpha Amylase in a Healthy Sample of Youth and Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Golda S. Ginsburg, Ph.D., Adjunct Professor, Johns Hopkins University
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: NA00083366; 1K24MH096760-01A1 (NIH)
Record Dates: First submitted 2015-07-01; First posted 2015-07-03 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-07

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Psychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Trier Social Stress Test (Experimental): Participants will be administered the Trier Social Stress Test (TSST). The TSST is the gold standard social stress test and involves speaking in front of confederate judges and completing arithmetic tasks. The task takes 10-15 minutes.
  Interventions: Behavioral: Trier Social Stress Test

INTERVENTIONS:
Behavioral: Trier Social Stress Test — The TSST is the gold standard social stress test and involves speaking in front of confederate judges and completing arithmetic tasks. The task takes 10-15 minutes.

SUMMARY:
The purpose of this study is to investigate how healthy youth and adults' cortisol levels and other hormone levels relate to anxiety levels while they participate in a behavioral task called the Trier Social Stress Task.

Data from these healthy participants will also be compared to those of anxious youth and adults collected as part of the in the Principal Investigator's ongoing study titled, "Child/Adolescent Anxiety Multimodal Extended Long-term Study (NA00035687)."

DETAILED DESCRIPTION:
The aim of this study is to investigate the independent and interactive associations linking salivary cortisol (a marker of hypothalamic-pituitary-adrenal activity or HPA activity) and alpha amylase (a marker of autonomic nervous system activity or ANS activity) in a sample of healthy controls. Data from these healthy controls will be compared in the future to clinically anxious youth. In this study, participants are asked to complete a one-time assessment consisting of interviews, questionnaires, and a behavioral task (called the Trier Social Stress Task) involving a short public speaking task and an arithmetic task in front of study staff. Throughout the behavioral task, study staff will collect four, small saliva samples using a straw-like tube from each participant. The assessment will take approximately 3 hours. Participants will be fully debriefed regarding the purposes of the stress procedure and assessed for any signs of residual distress. Since there is no treatment or randomization, blinding of study staff is not applicable. Participation in this study will not affect any current or future medical or psychiatric treatment.

AIMS: To examine whether a) salivary cortisol and alpha amylase response and recovery to the Trier Social Stress Task is associated with anxiety in non-psychiatrically ill participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant has no current psychiatric disorder
* Participant has no past psychiatric disorder
* Participant has no major medical disorder
* Participant is not currently receiving psychological or psychopharmacological treatment (medication) for any psychological disorder
* Participant is between the ages 11 and 34

Exclusion Criteria:

* Participant has or has had psychiatric disorder or medical condition contraindicating study participation
* Participant is pregnant
* Participant is not an English speaker
* Participant has a visual, motor, or hearing problem that would affect participation

Ages: 11 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2013-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Anxiety Disorders Interview Schedule for Diagnostic and Statistical Manual for Psychological Disorders-IV, Child and Parent Versions (C/P-ADIS), and Adult Versions (Client-ADIS) | 1 day
  The C/P and Client-ADIS' are semi-structured diagnostic interviews used to assess symptoms of anxiety, depression, and behavioral issues.
  This interview will be administered by a trained staff member and will utilize information from both parents and children (if child is under 18 years of age) or from the adult participant (if the participant is 18 years of age or older).
  This interview will be used to determine the presence or absence of an anxiety disorder for participants in this study.
  The ADIS is administered one time because each participant only completes a single study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Golda S Ginsburg, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States